CLINICAL TRIAL: NCT01949415
Title: An Optional Investigation of Biomarkers of Efficacy in TH002 Clinical Study Subjects.
Brief Title: An Optional Investigation of Biomarkers of Efficacy
Status: Completed | Type: Observational
Sponsor: Circassia Limited (Industry)
Collaborators: Adiga Life Sciences, Inc. (Industry); Topstone Research (Unknown)
Responsible Party: Sponsor
Other Study IDs: RES-008
Record Dates: First submitted 2013-09-20; First posted 2013-09-24 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Rhinoconjunctivitis
Keywords: House Dust Mite; Rhinoconjunctivitis; ToleroMune

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
House Dust Mites (HDM) are arachnids that infest bedding, carpet, upholstered furniture and fabric. Like many other allergens, exposure to HDMA in sensitised patients is associated with poorer lung function, greater medication requirements and more asthma symptoms as well as chronic rhinosinusitis symptoms. In contrast to other allergens, there is evidence that HDMA leads to the development of asthma, in addition to exacerbating pre-existing asthma in HDM-sensitised patients.

ToleroMune House Dust Mite (TM-HDM) is being developed for the treatment of HDM allergy.

Study TH002 evaluated the efficacy, safety and tolerability of TM-HDM. This study will identify cellular, proteomic or genetic biomarkers of efficacy to TM-HDM treatment in TH002 study participants

ELIGIBILITY:
Inclusion Criteria:

* Previously randomised into study TH002, completed the study and received either placebo or the 12 nmol dose in TH002.

Exclusion Criteria:

* Subjects who have received allergen or peptide immunotherapy during the last 12 months (other than TM-HDM)

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of subjects who completed TH002 and have been dosed with either placebo or the 12 nmol dose in the TH002 study.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
To identify cellular, proteomic or genetic biomarkers of efficacy to ToleroMune House Dust Mite (TM-HDM) treatment in TH002 study participants. | 1 Day

CONTACTS AND LOCATIONS:
Locations (1):
- Topstone Research, Toronto, Ontario, Canada